CLINICAL TRIAL: NCT07047001
Title: The Efficacy and Safety of Vorolanib Monotherapy or in Combination With Toripalimab for Postoperative Adjuvant Treatment of Renal Cell Carcinoma Patients With Intermediate-high Risk Recurrence Factors: A Multicenter, Randomized, Double-arm, Phase II Exploratory Study
Brief Title: Vorolanib Monotherapy or in Combination With Toripalimab as Adjuvant Therapy for Patients With Intermediate-high Risk of Recurrence in Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dong Wen (Other)
Responsible Party: Sponsor-Investigator, Dong Wen, chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-146-01
Record Dates: First submitted 2025-06-05; First posted 2025-07-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma (RCC); Adjuvant
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — vorolanib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- monotherpy (Experimental): Participants only received vorolanib as an adjuvant treatment.
  Interventions: Drug: Vorolanib Tablets
- combination therapy (Experimental): Participants received vorolanib combined with toripalimab as adjuvant therapy.
  Interventions: Drug: Vorolanib + Toripalimab

INTERVENTIONS:
Drug: Vorolanib Tablets — 200mg PO QD
  Other Names: CM082
  Arms: monotherpy
Drug: Vorolanib + Toripalimab — Vorolanib: 100mg PO QD
  Toripalimab: 240mg IV infusion Q3W
  Other Names: Toripalimab: JS001; Vorolanib:CM082
  Arms: combination therapy

SUMMARY:
While the 5-year survival rate for localized renal cell carcinoma (RCC) approaches 80%-95%, patients with high-risk non-metastatic disease face a substantial 30%-40% risk of recurrence/metastasis within 5 years. Emerging evidence demonstrates that combining anti-angiogenic agents with immune checkpoint inhibitors significantly extends progression-free survival (PFS) in first-line advanced/metastatic RCC settings. To address the unmet need for adjuvant strategies in intermediate/high-risk localized RCC, we propose a synergistic approach leveraging targeted therapy and immunotherapy. This dual-modality regimen may delay resistance mechanisms while enhancing disease-free survival (DFS) and overall survival (OS).

Vorolanib, a next-generation vascular endothelial growth factor receptor (VEGFR)-targeted tyrosine kinase inhibitor (TKI), exhibits unique pharmacodynamic properties that warrant investigation in adjuvant paradigms. This study evaluates two experimental arms: (1) Vorolanib combined with toripalimab, a PD-1 inhibitor. (2) Vorolanib monotherapy. This study aims to evaluate the efficacy and safety of vorolanib combined with toripalimab or vorolanib monotherapy in postoperative adjuvant therapy for intermediate/high-risk non-metastatic locally advanced renal cell carcinoma (RCC), while also investigating the correlation between postoperative minimal residual disease (MRD)-positive status and recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of localized and locally advanced stage renal cell carcinoma (RCC), with moderate to high recurrence risk
* Has intermediate-high risk, high risk, or M1 no evidence of disease (NED) RCC as defined by the following pathological tumor-node-metastasis and Fuhrman grading status:

  1. Intermediate-high risk RCC: pT1b-T2, Grade 4 or sarcomatoid, N0, M0; pT3, Any Grade, N0, M0;
  2. High risk RCC: pT4, Any Grade N0, M0; pT Any stage, Any Grade, N+, M0 M1 NED RCC participants who present not only with the primary kidney tumor but also solid, isolated, soft tissue metastases that can be completely resected at one of the following: the time of nephrectomy (synchronous) or, ≤1 year from nephrectomy (metachronous)
* Have adequate tissue for PD-L1 testing 0Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1
* Expected survival ≥ 12 months;
* Participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study treatment through 120 days after the last dose of study treatment
* Has adequate organ function
* Be able to understand and willing to sign the informed consent form

Exclusion Criteria:

* Patients with advanced/metastatic renal cell carcinoma (RCC) or non-clear cell renal cell carcinoma (nccRCC).
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies, or other agents specifically targeting T-cell co-stimulation checkpoints, or small molecule anti-angiogenic drugs.
* Subjects who underwent major surgery or chemotherapy within 4 weeks prior to the first dose administration, or those with postoperative duration >12 weeks who received major surgery/chemotherapy within 4 weeks before first dosing.
* Subjects with hypersensitivity to study drugs.
* Active hemorrhage, ulceration, intestinal perforation, bowel obstruction, or uncontrolled hypertension (defined as BP >140/90 mmHg or unstable during screening).
* Uncontrolled adrenal insufficiency.
* Congenital/acquired immunodeficiency (e.g., HIV infection) or active hepatitis:

HBV: HBsAg+ with HBV DNA ≥2000 IU/mL (≥10⁴ copies/mL) HCV: Anti-HCV+ with viral load >ULN

* Active autoimmune diseases (including but not limited to autoimmune hepatitis, interstitial lung disease, uveitis, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism) or history of autoimmune diseases. Exceptions: Vitiligo or childhood asthma fully resolved without intervention in adulthood.
* Symptomatic visceral metastases with imminent life-threatening complications (e.g., uncontrolled exudation [pleural/pericardial/abdominal], lymphangitic carcinomatosis, or >30% liver involvement).
* Severe infections requiring IV antibiotics/antifungals/antivirals within 4 weeks prior to first dose, or unexplained fever >38.5°C during screening.
* History of other malignancies within 5 years.
* Systemic corticosteroids or immunosuppressants within 14 days before first study drug administration.
* Documented active tuberculosis (Mycobacterium tuberculosis).
* Concurrent use of experimental agents or standard antineoplastic therapies.
* Active infections.
* High bleeding risk.
* Comorbidities (e.g., cardiopulmonary insufficiency) precluding radical nephrectomy/partial nephrectomy under general anesthesia.
* Pregnant/lactating women.
* Other conditions affecting trial conduct or interpretation (e.g., severe psychiatric disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
2-y DFS | From enrollment to the recurrence or metastasis or death(based on the first occurrence) at 2 years
  The proportion of patients who did not experience local recurrence/transfer or died for any reason within 2 years among all patients, per RECIST or irRECIST

SECONDARY OUTCOMES:
DFS | From date of enrollment until the date of local recurrence or distant metastasis occurs, or date of death from any cause ,whichever came first,assessed up to 100 months
  The period from the date of enrollment until local recurrence or distant metastasis occurs, or until death due to any cause, shall be measured from the earlier of the two events, per RECIST 1.1 and irRECIST
OS | From date of enrollment to death due to any cause,assessed up to 120 months
  The period from the date of enrollment until the date of death due to any cause
Safety and tolerability | 1 year
  The proportion of patients experiencing adverse events among the total patients, per CTCEA v5.0
The correlation between MRD positivity and recurrence | up to 2 years
  The correlation between postoperative MRD (Minimal Residual Disease) positive status and postoperative recurrence
Correlation between molecular characteristics and therapeutic efficacy | up to 2 years
  Calculate the MRD positive rate of the patients.All of the patients were divided into negative group and positive group based on the MRD status.Evaluate the RFS of the two groups separately, and the evaluation index was the hazard ratio（HR）value.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China